CLINICAL TRIAL: NCT03950128
Title: Healthy Relationships Training Study: Comparing the Efficacy of a Mindfulness-Based Skills Training to a Psychoeducational Intervention at Reducing Dating Violence on College Campuses
Brief Title: Healthy Relationships Training Study: A Comparison of Interventions to Reduce Dating Violence on College Campuses
Acronym: HRTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Manfred van Dulmen, Associate Dean, Professor of Psychological Sciences, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-547
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Dating Violence
Keywords: Dating aggression; Emotion regulation; Mindfulness; Mindfulness-based skills; Romantic relationships; Dating relationships
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Skills Training (Experimental): This intervention teaches students mindfulness-based skills to help manage their emotions when resolving conflict with their partners. The intervention is given over the course of three 50-minute sessions with homework between sessions.
  Interventions: Behavioral: Mindfulness-Based Skills Training (MBST)
- Psychoeducational (Active Comparator): This intervention is based on the Love is Not Abuse (LINA) Curriculum (Liz Claiborne Education Development Center (n.d.)). It was adapted to be given over the course of three 50-minute sessions.
  Interventions: Behavioral: Psychoeducational

INTERVENTIONS:
Behavioral: Mindfulness-Based Skills Training (MBST) — This intervention teaches students mindfulness-based skills to help manage their emotions when resolving conflict with their partners. The skills followed the "ABCDE" acronym. ABCDE stands for awareness, breathing, checking in with your feelings and thoughts, describing your experience, and expressing what you want to change. Students learned about the skills and had opportunities to practice them as well.
  Arms: Mindfulness-Based Skills Training
Behavioral: Psychoeducational — This intervention is based on the Love is Not Abuse (LINA) Curriculum (Liz Claiborne Education Development Center (n.d.)). It was adapted to be given over the course of three 50-minute sessions. The selected materials covered (a) what dating abuse is, (b) the pattern of abuse and, (c) technology and dating abuse. The curriculum is interactive and includes handouts, activities, and discussion.
  Arms: Psychoeducational

SUMMARY:
The purpose of this study is to compare the efficacy of a mindfulness-based skills training (MBST) to a psychoeducational intervention at reducing dating violence in a sample of college students. The MBST focuses on improving college students' abilities to manage emotionally charged states during conflict with their romantic partners by teaching them mindfulness-based skills. The psychoeducational intervention uses the Love is Not Abuse curriculum. Treatment groups are randomly assigned and are compared using a two-armed parallel design.

88 college students currently in a dating relationship were recruited through Kent State University's subject pool. All participants completed a baseline assessment online where self-reported data was collected on demographics, dating violence (during the past month), emotion regulation, mindfulness skills, and other potential covariates. Participants were then randomized into either the MBST intervention or the psychoeducational intervention. All participants completed three 50-minute sessions over the course of three weeks with assigned homework between sessions. Daily diary data was collected, assessing knowledge and use of skills learned in the sessions. Follow-up data was collected online 11 weeks following baseline (dating violence (during the last month), emotion regulation, mindfulness skills).

It was hypothesized that the MBST intervention would be more effective at reducing dating violence as compared to the psychoeducational intervention.

ELIGIBILITY:
Inclusion Criteria:

* In a current dating relationship (of 6 months or longer)

Exclusion Criteria:

* Diagnosed with psychopathology (Major Depressive Disorder, Post-Traumatic Stress Disorder, Borderline Personality Disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Conflict in Adolescent Dating Relationships Inventory (CADR; Wolfe et al., 2001) | Baseline (4th week of semester) and Follow-up (11 weeks after baseline)
  A 35-item self-report measure of physical, verbal, and sexual dating violence.

SECONDARY OUTCOMES:
Kentucky Inventory of Mindfulness Skills (KIMS; Baer, Smith, & Allen, 2004) | Baseline (4th week of semester) and Follow-up (11 weeks after baseline)
  This self-report measure has a total of 39 items with four subscales that assess: observing (e.g., I notice when my moods begin to change), describing (e.g., I'm good at finding the words to describe my feelings), accepting without judgment (e.g., I criticize myself for having irrational or inappropriate emotions [reverse scored]), and acting with awareness (e.g., When I'm doing something, I'm only focused on what I'm doing, nothing else).
The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Baseline (4th week of semester) and Follow-up (11 weeks after baseline)
  This self-report measure asks participants to indicate how often a series of items applies to them (36 items total), rated on a 5-point scale (1 = almost never, 2 = sometimes, 3 = about half of the time, 4 = most of the time, 5 = almost always). The six subscales are: lack of emotional awareness (e.g., "When I'm upset, I take time to figure out what I'm really feeling" [reverse scored]), lack of emotional clarity (e.g., "I have difficulty making sense out of my feelings"), nonacceptance of emotional responses (e.g., "When I'm upset, I become angry with myself for feeling that way"), impulse control difficulties (e.g., "When I'm upset, I lose control over my behaviors"), limited access to emotion regulation strategies (e.g., "When I'm upset, believe that wallowing in it is all I can do"), and difficulties engaging in goal-directed behavior (e.g., "When I'm upset, I have difficulty thinking about anything else").
3. Intimate Partner Violence Attitudes Scale-Revised (IPVAS-R; Fincham, Cui, Braithwaite, & Pasley, 2008) | Baseline (4th week of semester) and Follow-up (11 weeks after baseline)
  This self-report measure asks participants to indicate how strongly they agree or disagree with a series of 17 statements on a five-point Likert scale (1 = Strongly disagree, 5 = Strongly agree). There are three subscales: abuse (e.g., "During a heated argument, it is okay for me to bring up something from my partner's past to hurt him or her"), control (e.g., "It is okay for me to tell my partner not to talk to someone of the opposite sex"), and violence (e.g., "It would never be appropriate to hit or try to hit one's partner with an object" [reverse scored]).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred van Dulmen, PhD, Principal Investigator — Kent State University
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The PI and co-PI are the only researchers involved in the project. Thus, no plans for sharing are necessary.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03950128/Prot_SAP_000.pdf